CLINICAL TRIAL: NCT06458309
Title: Management of Spine Fractures According to The Thoracolumbar AO Spine Injury Score
Brief Title: Mangement of Spine Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Youssef Rady Youssef, Resident- orthopedic department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh_med_24_05_04ms
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Spine Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spine surgery — AO Classification6 It classifies thoracolumbar fractures into 3 major groups, based on the mechanism of injury.and each of them subdivided to 3 subgroups.
  A. Compression B. Distraction C. multi-directional with translation Thoracolumbar AO spine injury score

SUMMARY:
Each year, there are approximately 5 million new vertebral fractures worldwide1. Most of these fractures involve the thoracolumbar or lumbar spines. The thoracolumbar junction, due to its mechanical transition zone, and the lumbar spine, due to its absence of stabilizing articulations with the ribs, lordotic posture and more sagittal oriented facet joints, are vulnerable for involvement in spinal injuries2.

Burst fractures occurs frequently in high-energy traumas which are most commonly associated with falls and traffic accidents.3

ELIGIBILITY:
Inclusion Criteria:

* 1-Skeletally mature patients (18yrs and older). 2-Thoracolumbar fractures.

Exclusion Criteria:

* 1-skeletally immature patients. 2-pathological fractures.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
AO Spine Injury Score | 1 year
  * injury morphology
  * integrity of the PLC
  * neurological status

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hu R, Mustard CA, Burns C. Epidemiology of incident spinal fracture in a complete population. Spine (Phila Pa 1976). 1996 Feb 15;21(4):492-9. doi: 10.1097/00007632-199602150-00016. PMID 8658254
- [Background] Tran NT, Watson NA, Tencer AF, Ching RP, Anderson PA. Mechanism of the burst fracture in the thoracolumbar spine. The effect of loading rate. Spine (Phila Pa 1976). 1995 Sep 15;20(18):1984-8. doi: 10.1097/00007632-199509150-00004. PMID 8578372
- [Background] Bohlman HH. Treatment of fractures and dislocations of the thoracic and lumbar spine. J Bone Joint Surg Am. 1985 Jan;67(1):165-9. No abstract available. PMID 3881446
- [Background] McAfee PC, Yuan HA, Fredrickson BE, Lubicky JP. The value of computed tomography in thoracolumbar fractures. An analysis of one hundred consecutive cases and a new classification. J Bone Joint Surg Am. 1983 Apr;65(4):461-73. PMID 6833320